CLINICAL TRIAL: NCT03244735
Title: Efficacy of Modified Atkins Ketogenic Diet in Chronic Cluster Headache. A Prospective Case Series
Brief Title: Efficacy of Modified Atkins Ketogenic Diet in Chronic Cluster Headache: a Prospective Case Series
Acronym: CCHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Cherubino DI LORENZO, Research Fellow, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHDiet
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Chronic Cluster Headache
Keywords: Ketogenic Diet
MeSH Terms: conditions — Cluster Headache | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Atkins Diet (MAD) (Experimental): CCH patients that follows at least 3 months of MAD
  Interventions: Other: Atkins diet

INTERVENTIONS:
Other: Atkins diet — A nutritional regimen characterized by high fat low carbohydrate intake.

SUMMARY:
Atkins diet is a nutritional regimen characterized by ad libitum protein and fat intake, but carbohydrate restriction. It is followed by millions of people around the word as a life-style, but in the last years was proposed as a treatment for the epilepsy, by its capacity to induce the state of ketosis.

Since Authors observed that ketosis could be also useful in migraine, and migraine shares some pathophysiological features with cluster headache, The aim of the study is to test the efficacy of Atkins diet in Cluster Headache by an open label one harm observational study.

DETAILED DESCRIPTION:
The Atkins diet is a ketogenic high-fat, low-carbohydrate diet for long adopted as lifestyle by people that dislike have an high carbohydrate intake. This nutritional life style seems to account for more energy in the daily activity and an easy weight control. In the last years, researchers showed that a modified Atkins diet (MAD) can be useful to treat drug resistant epilepsy, maybe by the induction of ketogenesis.

Ketogenesis, ketone-body formation, is a physiologic phenomenon also observed in patients following low-carbohydrate high fat diets. Different Authors evidenced a protective effect of ketone bodies also on migraine that shares some pathophysiological features with cluster headache (CH).

CH is the worst form of headache, also called as "suicide headache"; in particular its unremitting form, called Chronic CH (CCH) is regarded as a clinical challenge for neurologist, if refractory to pharmacological treatments. So far, no data are available about a beneficial effect of ketogenesis in CH. However, the beta hydroxybutyrate (BHB) has a chemical formula similar to gamma hydroxybutyrate (GHB) that has shown to be effective in CH. Moreover, ketosis has also a beneficial effect on hypothalamic dysfunctions that are shared by some form of epilepsy and CH.

Aim of this study is verify in an open label observational study if a MAD can be useful in the treatment of CCH. In case of positive outcome, the results could be used as preliminary data to design a double blind versus placebo study, to asses definitively if ketogenesis is really able to prevent/avoid headache attacks in CH.

Methods: By the Italian branch of the Organization for the Understanding of Cluster Headache (OUCH), there will be recruited CCH volunteers that accept to modify their diet according to Atkins Diet for at least three months.

Headache attack frequency will be collected on specific headache-calendars and a comparison between the pre-diet phase and the during-the-diet- phase will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CCH (less than 30 consecutive days of attacks remission in the last year)
* kept a headache diary for at least 1 month
* CH onset before the age of 50

Exclusion Criteria:

* over consumption of acute pain-killers (triptan, analgesic, or ergotamine)
* pregnancy or lactation
* type I diabetes
* serious organic or psychiatric disorders that the investigators judged as having the potential to influence the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Attack frequency | 3 months
  Reduction of at least 50% of number of attacks per month

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pierelli, MD, Study Chair — Sapienza Univeristy
Locations (1):
- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
We do not share data

REFERENCES:
- [Background] Di Lorenzo C, Coppola G, Sirianni G, Rossi P, Pierelli F. O045. Cluster headache improvement during Ketogenic Diet. J Headache Pain. 2015 Dec;16(Suppl 1):A99. doi: 10.1186/1129-2377-16-S1-A99. No abstract available. PMID 28132289
- [Derived] Di Lorenzo C, Coppola G, Di Lenola D, Evangelista M, Sirianni G, Rossi P, Di Lorenzo G, Serrao M, Pierelli F. Efficacy of Modified Atkins Ketogenic Diet in Chronic Cluster Headache: An Open-Label, Single-Arm, Clinical Trial. Front Neurol. 2018 Feb 12;9:64. doi: 10.3389/fneur.2018.00064. eCollection 2018. PMID 29483892